CLINICAL TRIAL: NCT03398408
Title: Cognitive Flexibility Training in Persistent Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Lumos Labs, Inc. (Industry)
Responsible Party: Principal Investigator, simon.haroutounian, Assistant Professor of Anesthesiology, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 201706064
Record Dates: First submitted 2017-12-28; First posted 2018-01-12 (Actual); Last update posted 2020-05-06 (Actual); Status verified 2020-05

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Patients in both groups will complete paper-pencil TMT A and B and the CWMST, the computer-based TMT A and B and Color Match, and NCPT tests upon enrollment into the study.
  Participants in the intervention group will then be provided with the Lumosity cognitive flexibility training module and complete daily training for a total of five weeks. 1-3 days after completion of their training, all patients will be invited to complete the computerized versions of the TMT A and B, Color Match, and NCPT tests again on their personal computers.
  Interventions: Behavioral: Training
- Control (No Intervention): Patients in both groups will complete paper-pencil TMT A and B and the CWMST, the computer-based TMT A and B and Color Match, and NCPT tests upon enrollment into the study.
  Patients in the control group will complete all tests upon enrollment and approximately five weeks after their initial testing, but will not participate in training.

INTERVENTIONS:
Behavioral: Training — The intervention group will be provided with the cognitive training module and participants will be required to complete a targeted 36-minute daily training for 35 days.
  Arms: Intervention

SUMMARY:
To determine whether participation in a cognitive training program over a training period of five weeks improves cognitive flexibility in patients with chronic hip, knee, and back pain.

DETAILED DESCRIPTION:
This project is a single-center prospective, randomized study to assess whether cognitive flexibility can be improved through training on a Lumosity®-based training module over the course a five week timeframe in patients with chronic hip, knee, and back pain; and whether changes in cognitive flexibility will correlate with perceived pain scores.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 18 to 70 with chronic hip, knee, or low back pain for >3 months
* Documented moderate to severe chronic pain
* English as a primary language
* Access to a computer at home and an email account

Exclusion Criteria:

* Diagnosed Alzheimer's or documented severe cognitive impairment
* Lack of email/lack of basic computer skills
* Has undergone an interventional pain procedure within one week prior to enrollment
* Are scheduled to undergo a pain procedure during the five weeks of complete cognitive training

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2017-12-29 (Actual); Primary Completion 2019-08-07 (Actual); Study Completion 2019-08-07 (Actual)

PRIMARY OUTCOMES:
Does cognitive training over five weeks improve cognitive flexibility performance scores in chronic hip, knee, and back pain patients? | Up to 5 months
  The primary outcome, i.e. NCPT score, will be assessed before and after five weeks of cognitive training. T-test will be used to compare the change in NCPT score between the training and the control group.

CONTACTS AND LOCATIONS:
Overall Officials: Simon Haroutounian, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University in St. Louis, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
ADD

REFERENCES:
- [Background] Kehlet H, Jensen TS, Woolf CJ. Persistent postsurgical pain: risk factors and prevention. Lancet. 2006 May 13;367(9522):1618-25. doi: 10.1016/S0140-6736(06)68700-X. PMID 16698416
- [Background] Haroutiunian S, Nikolajsen L, Finnerup NB, Jensen TS. The neuropathic component in persistent postsurgical pain: a systematic literature review. Pain. 2013 Jan;154(1):95-102. doi: 10.1016/j.pain.2012.09.010. PMID 23273105
- [Background] Smith BH, Torrance N. Epidemiology of neuropathic pain and its impact on quality of life. Curr Pain Headache Rep. 2012 Jun;16(3):191-8. doi: 10.1007/s11916-012-0256-0. PMID 22395856
- [Background] Dworkin RH, Panarites CJ, Armstrong EP, Malone DC, Pham SV. Healthcare utilization in people with postherpetic neuralgia and painful diabetic peripheral neuropathy. J Am Geriatr Soc. 2011 May;59(5):827-36. doi: 10.1111/j.1532-5415.2011.03403.x. PMID 21568954
- [Background] Clarke H, Soneji N, Ko DT, Yun L, Wijeysundera DN. Rates and risk factors for prolonged opioid use after major surgery: population based cohort study. BMJ. 2014 Feb 11;348:g1251. doi: 10.1136/bmj.g1251. PMID 24519537
- [Background] Apfelbaum JL, Chen C, Mehta SS, Gan TJ. Postoperative pain experience: results from a national survey suggest postoperative pain continues to be undermanaged. Anesth Analg. 2003 Aug;97(2):534-540. doi: 10.1213/01.ANE.0000068822.10113.9E. PMID 12873949
- [Background] Oosterman JM, Dijkerman HC, Kessels RP, Scherder EJ. A unique association between cognitive inhibition and pain sensitivity in healthy participants. Eur J Pain. 2010 Nov;14(10):1046-50. doi: 10.1016/j.ejpain.2010.04.004. Epub 2010 May 20. PMID 20493746
- [Background] Baliki MN, Mansour AR, Baria AT, Apkarian AV. Functional reorganization of the default mode network across chronic pain conditions. PLoS One. 2014 Sep 2;9(9):e106133. doi: 10.1371/journal.pone.0106133. eCollection 2014. PMID 25180885
- [Background] Kucyi A, Salomons TV, Davis KD. Cognitive behavioral training reverses the effect of pain exposure on brain network activity. Pain. 2016 Sep;157(9):1895-1904. doi: 10.1097/j.pain.0000000000000592. PMID 27101426
- [Background] Vachon-Presseau E, Tetreault P, Petre B, Huang L, Berger SE, Torbey S, Baria AT, Mansour AR, Hashmi JA, Griffith JW, Comasco E, Schnitzer TJ, Baliki MN, Apkarian AV. Corticolimbic anatomical characteristics predetermine risk for chronic pain. Brain. 2016 Jul;139(Pt 7):1958-70. doi: 10.1093/brain/aww100. Epub 2016 May 5. PMID 27190016
- [Background] Lamm C, Decety J, Singer T. Meta-analytic evidence for common and distinct neural networks associated with directly experienced pain and empathy for pain. Neuroimage. 2011 Feb 1;54(3):2492-502. doi: 10.1016/j.neuroimage.2010.10.014. Epub 2010 Oct 12. PMID 20946964
- [Background] Bernardy K, Klose P, Busch AJ, Choy EH, Hauser W. Cognitive behavioural therapies for fibromyalgia. Cochrane Database Syst Rev. 2013 Sep 10;2013(9):CD009796. doi: 10.1002/14651858.CD009796.pub2. PMID 24018611
- [Background] Attal N, Masselin-Dubois A, Martinez V, Jayr C, Albi A, Fermanian J, Bouhassira D, Baudic S. Does cognitive functioning predict chronic pain? Results from a prospective surgical cohort. Brain. 2014 Mar;137(Pt 3):904-17. doi: 10.1093/brain/awt354. Epub 2014 Jan 17. PMID 24441173
- [Background] Bowie CR, Harvey PD. Administration and interpretation of the Trail Making Test. Nat Protoc. 2006;1(5):2277-81. doi: 10.1038/nprot.2006.390. PMID 17406468
- [Background] Kortte KB, Horner MD, Windham WK. The trail making test, part B: cognitive flexibility or ability to maintain set? Appl Neuropsychol. 2002;9(2):106-9. doi: 10.1207/S15324826AN0902_5. PMID 12214820
- [Background] Uttl B, Graf P. Color-Word Stroop test performance across the adult life span. J Clin Exp Neuropsychol. 1997 Jun;19(3):405-20. doi: 10.1080/01688639708403869. PMID 9268815
- [Background] Morrison GE, Simone CM, Ng NF, Hardy JL. Reliability and validity of the NeuroCognitive Performance Test, a web-based neuropsychological assessment. Front Psychol. 2015 Nov 3;6:1652. doi: 10.3389/fpsyg.2015.01652. eCollection 2015. PMID 26579035
- [Background] Tombaugh TN. Trail Making Test A and B: normative data stratified by age and education. Arch Clin Neuropsychol. 2004 Mar;19(2):203-14. doi: 10.1016/S0887-6177(03)00039-8. PMID 15010086
- See also: IASP Task Force for the Classification of Chronic Pain in ICD-11 Prepares New Criteria on Postsurgical and Posttraumatic Pain — https://www.iasp-pain.org/PublicationsNews/NewsDetail.aspx?ItemNumber=5134&navItemNumber=643